CLINICAL TRIAL: NCT00362323
Title: A Randomized, Double-blind Study Comparing the Efficacy and Safety of a Fixed Combination of Fenofibrate and Metformin vs Metformin Alone in Patients With Type 2 Diabetes Mellitus and Dyslipidemia Not Appropriately Controlled With a Statin.
Brief Title: Fenofibrate and Metformin Fixed Combination vs Metformin - FAME METFO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C LF23-0121 06 01; 2006-000924-15
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Dyslipidemia/Glucose Metabolism Disorder
Keywords: Treatment of Dyslipidemia and of Type 2 Diabetes Mellitus
MeSH Terms: conditions — Dyslipidemias; Glucose Metabolism Disorders | interventions — Fenofibrate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: fenofibrate (F) + metformin (M) hydrochloride fixed combination
- 2 (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: fenofibrate (F) + metformin (M) hydrochloride fixed combination — F80mg/M500mg - per os - twice a day during 24 weeks / or / F80mg/M850mg - per os - twice a day during 24 weeks /or / F54mg/M850mg - per os - three times a day during 24 weeks
  Arms: 1
Drug: Metformin — 500mg - per os - twice a day during 24 weeks /or / 850mg - per os - twice a day during 24 weeks /or / 850mg - per os - three times a day during 24 weeks
  Arms: 2

SUMMARY:
To demonstrate in patients with T2DM and dyslipidemia not appropriately controlled with a statin and receiving metformin, the superiority of a fixed combination of fenofibrate and metformin vs metformin alone on TG and additionally, if the superiority on TG is established, to demonstrate the superiority on HDL-C

ELIGIBILITY:
Inclusion Criteria Patient with Type 2 Diabetes treated with stable dose of metformin and with dyslipidemia not appropriately controlled with a statin treatment.

Exclusion Criteria Type 1 diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
TG / HDL-C ratio | 24 weeks

SECONDARY OUTCOMES:
Lipid and glycemic parameters | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michel Conte, Study Director — Solvay Pharmaceuticals
Locations (70):
- Czechia (9):
  - C LF23-0121 06 01 Site107, Brno
  - C LF23-0121 06 01 Site108, Holešov
  - C LF23-0121 06 01 Site101, Karlovy Vary
  - C LF23-0121 06 01 Site106, Olomouc
  - C LF23-0121 06 01 Site109, Olomouc
  - C LF23-0121 06 01 Site103, Pardubice
  - C LF23-0121 06 01 Site102, Prague
  - C LF23-0121 06 01 Site104, Prague
  - C LF23-0121 06 01 Site105, Prague
- France (7):
  - C LF23-0121 06 01 Site 204, Bailleul
  - C LF23-0121 06 01 Site 200, Bondy
  - C LF23-0121 06 01 Site 207, Cholet
  - C LF23-0121 06 01 Site 208, Évreux
  - C LF23-0121 06 01 Site 201, Pantin
  - C LF23-0121 06 01 Site 202, Tours
  - C LF23-0121 06 01 Site 205, Wattrelos
- Hungary (9):
  - C LF23-0121 06 01 Site 406, Balatonfüred
  - C LF23-0121 06 01 Site 400, Budapest
  - C LF23-0121 06 01 Site 401, Budapest
  - C LF23-0121 06 01 Site 402, Budapest
  - C LF23-0121 06 01 Site 403, Budapest
  - C LF23-0121 06 01 Site 405, Budapest
  - C LF23-0121 06 01 Site 407, Budapest
  - C LF23-0121 06 01 Site 408, Budapest
  - C LF23-0121 06 01 Site 404, Debrecen
- India (16):
  - C LF23-0121 06 01 Site 501, Bangalore
  - C LF23-0121 06 01 Site 504, Bangalore
  - C LF23-0121 06 01 Site 516, Bangalore
  - C LF23-0121 06 01 Site 519, Bangalore
  - C LF23-0121 06 01 Site 508, Chennai
  - C LF23-0121 06 01 Site 510, Chennai
  - C LF23-0121 06 01 Site 505, Hyderabad
  - C LF23-0121 06 01 Site 509, Hyderabad
  - C LF23-0121 06 01 Site 517, Hyderabad
  - C LF23-0121 06 01 Site 511, Karnataka
  - C LF23-0121 06 01 Site 512, Maharashtra
  - C LF23-0121 06 01 Site 502, Mumbai
  - C LF23-0121 06 01 Site 503, Mumbai
  - C LF23-0121 06 01 Site 518, Nashik
  - C LF23-0121 06 01 Site 506, Pune
  - C LF23-0121 06 01 Site 514, Tiruvanathapuram-Kerala
- Lithuania (3):
  - C LF23-0121 06 01 Site 800, Vilnius
  - C LF23-0121 06 01 Site 801, Vilnius
  - C LF23-0121 06 01 Site 802, Vilnius
- Poland (22):
  - C LF23-0121 06 01 Site 600, Bialystok
  - C LF23-0121 06 01 Site 613, Bydgoszcz
  - C LF23-0121 06 01 Site 618, Grudziądz
  - C LF23-0121 06 01 Site 603, Katowice
  - C LF23-0121 06 01 Site 601, Krakow
  - C LF23-0121 06 01 Site 607, Krakow
  - C LF23-0121 06 01 Site 610, Krakow
  - C LF23-0121 06 01 Site 615, Kutno
  - C LF23-0121 06 01 Site 605, Olsztyn
  - C LF23-0121 06 01 Site 604, Opole
  - C LF23-0121 06 01 Site 606, Poznan
  - C LF23-0121 06 01 Site 609, Poznan
  - C LF23-0121 06 01 Site 621, Sliwinska
  - C LF23-0121 06 01 Site 617, Starogard Gdański
  - C LF23-0121 06 01 Site 616, Szczecin
  - C LF23-0121 06 01 Site 602, Warsaw
  - C LF23-0121 06 01 Site 608, Warsaw
  - C LF23-0121 06 01 Site 619, Warsaw
  - C LF23-0121 06 01 Site 620, Warsaw
  - C LF23-0121 06 01 Site 611, Wroclaw
  - C LF23-0121 06 01 Site 612, Wroclaw
  - C LF23-0121 06 01 Site 614, Zgierz
- Slovakia (4):
  - C LF23-0121 06 01 Site 700, Bratislava
  - C LF23-0121 06 01 Site 703, Košice
  - C LF23-0121 06 01 Site 702, Lučenec
  - C LF23-0121 06 01 Site 701, Skalica